CLINICAL TRIAL: NCT02110719
Title: Decreasing Narcotics in Advanced Pelvic Surgery: A Randomized Study
Brief Title: Decreasing Narcotics in Advanced Pelvic Surgery
Acronym: Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REAG00414HU
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Narcotic Use; Pain; Constipation; Nausea
Keywords: narcotic use; pain; constipation; nausea
MeSH Terms: conditions — Pain; Constipation; Nausea | interventions — Celecoxib; Gabapentin; Acetaminophen; Ibuprofen; oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination; Oxycodone; Hydromorphone; Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Patients will be given the following:
  * no preoperative medications
  * intraoperative medications per anesthesia
  * postoperatively, patients will receive ibuprofen, tylenol and narcotics as needed
  Interventions: Drug: oral acetaminophen; Drug: oral ibuprofen; Drug: percocet; Drug: vicodin; Drug: dilaudid
- Multimodal (Active Comparator): Patients in the multimodal arm will receive the following:
  * preoperative celebrex and gabapentin
  * intraoperative IV acetaminophen, dexamethasone, zofran
  * postoperative scheduled IV acetaminophen, PO celebrex and gabapentin, and as needed PO narcotics
  * patient will be discharged on scheduled ibuprofen and acetaminophen for 3 days followed by "as needed" use as well as "as needed" narcotics
  Interventions: Drug: Celebrex; Drug: Gabapentin; Drug: IV acetaminophen; Drug: oral acetaminophen; Drug: oral ibuprofen; Drug: Oxycodone; Drug: dilaudid; Drug: Dexamethasone; Drug: zofran

INTERVENTIONS:
Drug: Celebrex
  Arms: Multimodal
Drug: Gabapentin
  Arms: Multimodal
Drug: IV acetaminophen
  Arms: Multimodal
Drug: oral acetaminophen
Drug: oral ibuprofen
Drug: percocet
  Arms: Standard
Drug: vicodin
  Arms: Standard
Drug: Oxycodone
  Arms: Multimodal
Drug: dilaudid
Drug: Dexamethasone
  Arms: Multimodal
Drug: zofran
  Arms: Multimodal

SUMMARY:
In recent years, there has been an emphasis on the creation of "enhanced-recovery", "fast-track" or "multi-modal" pathways to improve perioperative care (1-4). The goal of these programs is to reduce the length of hospital stay, decrease narcotic usage while improving pain control, accelerate post-operative recovery, and expedite return to baseline functional status. Pathways often are developed by a team of surgeons, nurses, pain specialists, anesthesiologists and other support staff. Postoperative components often involve multi-modal analgesia, early return to activity and early return to a regular diet. The goal of this study is to evaluate the efficacy of a multi-modal pain regimen in advanced pelvic surgery with a primary goal of decreasing narcotic usage.

ELIGIBILITY:
Inclusion Criteria:

* women >/= 18 years old
* undergoing pelvic organ prolapse or incontinence surgery with the Urogynecology department

Exclusion Criteria:

* males
* <18 years old
* women unwilling or unable to consent
* same-day-discharge surgery
* history of chronic pain for which they use medications
* current or active history of narcotic abuse
* sleep apnea
* liver or kidney dysfunction
* sulfa allergy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Narcotic use | intraoperative, immediate postoperative and 1 week postoperative
  Narcotic use will be evaluated at all stages of the preoperative care: operating room, hospital floor and at the 1 week postoperative time point

SECONDARY OUTCOMES:
Pain | postoperative day #1 and postoperative week #1
  pain will be evaluated at the above listed time points using the validated brief pain inventory
Nausea | intraoperatively, postoperatively
  Nausea will be evaluated based on the use of narcotics in the hospital
Constipation | one week postoperatively
  constipation at the time of the first bowel movement will be evaluated using the validated Bristol Stool Scale

CONTACTS AND LOCATIONS:
Overall Officials: Krista Reagan, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hosptial, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No